CLINICAL TRIAL: NCT06534138
Title: An Observational Study on the Role of Exercise in the Disease Progression of Chronic Pancreatitis.
Brief Title: Exercise Inhibit Innate Immune Response and Ameliorate Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Exercise
Record Dates: First submitted 2024-03-25; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-Chronic Pancreatitis (Non-CP): Patients diagnosed without chronic pancreatitis based on imaging results were categorized into the Non-CP group.
- Chronic Pancreatitis-non-exercise (CP-non-exercise): Patients diagnosed with chronic pancreatitis based on imaging results, while simultaneously not engaging in physical exercise, were categorized into the CP-non-exercise group.
- Chronic Pancreatitis-exercise (CP-exercise): Patients diagnosed with chronic pancreatitis based on imaging results, while concurrently adhering to physical exercise, were categorized into the CP-exercise group.
  Interventions: Behavioral: Physical exercise

INTERVENTIONS:
Behavioral: Physical exercise — The CP-exercise group was categorized based on patients' self-reported daily exercise time into four levels: 15 minutes/day, 30 minutes/day, 45 minutes/day, and ≥60 minutes/day. Additionally, resistance exercise and endurance exercise were distinguished based on patients' self-reported exercise modalities, including swimming, jogging, brisk walking, practicing Tai Chi, and dumbbell training.
  Groups: Chronic Pancreatitis-exercise (CP-exercise)

SUMMARY:
The goal of this observational study is to learn about the effects of different physical exercise on disease progression in patients with chronic pancreatitis. The main question it aims to answer is:

Can physical exercise alleviate the disease progression of chronic pancreatitis?

Currently, the investigators have followed up with participants through a telephone questionnaire for six months to investigate whether the participants have engaged in physical exercise and to assess the disease progression of chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic pancreatitis
* Must be adhere to the guidelines of the American Gastroenterological Association

Exclusion Criteria:

* Autoimmune pancreatitis
* Pancreatic cancer diagnosed within 2 years after the onset of CP
* Use of drugs or toxins, or presence of viral infections

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The 105 patients with CP were categorized into the sedentary group (CP-Sed, n = 54) and exercise group (CP-Ex, n = 51) based on self-reported exercise time per day during the six-month follow-up post the diagnosis of CP. Physical exercise time was recorded at four levels: 15 min/d, 30 min/d, 45 min/d, and 60 min/d or more.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Physical Exercise Can Alleviate the Disease Progression of Chronic Pancreatitis. | Six months
  The investigators collected data on patients' exercise time and modalities through telephone questionnaires. The impact of exercise on patients with chronic pancreatitis was determined by assessing VAS scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China